CLINICAL TRIAL: NCT04631575
Title: A Single Dose, Open-label, Parallel Controlled Pharmacokinetic Study of SHR6390 in Participants With Mild to Moderate Liver Impairment and Healthy Participants
Brief Title: An Investigational Study of SHR6390 in Participants With Mild to Moderate Liver Impairment and Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHR6390-I-109
Record Dates: First submitted 2020-11-13; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Hepatic Impairment; Healthy Participants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy participants (Experimental): Intervention: Drug: SHR6390 single dose
  Interventions: Drug: SHR6390
- Mild liver impairment (Experimental): Intervention: Drug: SHR6390 single dose
  Interventions: Drug: SHR6390
- Moderate liver impairment (Experimental): Intervention: Drug: SHR6390 single dose
  Interventions: Drug: SHR6390

INTERVENTIONS:
Drug: SHR6390 — SHR6390, PO,single-dose

SUMMARY:
The purpose of this study is to investigate SHR6390 in participants with different levels of liver function

ELIGIBILITY:
Inclusion Criteria:

-

Participants with mild to moderate liver impairment must meet all of the following criteria to enter the study:

* The informed consent is signed before the trial, and the content, process and possible adverse reactions are fully understood; Be able to complete the study according to the requirements of the test scheme;
* Both male and female, subjects aged 18 to 65 years (including both ends) on the date of signing informed consent;
* The body weight of male subjects is ≥50 kg, while female subjects is ≥45 kg. Body mass index (BMI) is in the range of 18.5 kg/m2-30 kg/m2;
* Chronic stable primary liver disease is necessary for patients with liver impairment, then patients with Grade-A/mild liver impairment (Child-Pugh score: 5-6) and Grade-B/moderate liver impairment (Child-Pugh score: 7-6) are assessed according to Child-Pugh classification;
* Provide documentary evidence of confirmed liver impairment;
* Patients who have stable medication regimen for liver impairment, complications and other concomitant diseases within at least 28 days before taking the experimental drug, and the medication does not need to be adjusted (including drug type, dosage or frequency) during the clinical trials; or those who do not use the drug;
* The function of vital organs meets the following criteria: Absolute neutrophil count (ANC) ≥ 1.0 × 109 / L (1000 / mm3); Platelet ≥ 75.0 × 109 / L (75000 / mm3); Hemoglobin (Hgb) ≥ 9.0 g / dL (90g / L); ALT and AST ≤ 5ULN; Creatinine clearance rate (CLcr) ≥ 60 mL / min; The corrected QTc interval (QTcF) ≤ 450 msec (male), ≤ 470 msec (female);
* In addition to liver impairment and complications, the investigator judged good condition according to the history inquiry, vital signs, physical examination, routine laboratory examination, 12-lead ECG, EEG, etc., and there was no other clinically significant abnormality;
* No family planning during the trial and within 6 months after the last administration of the trial drug, and voluntarily take effective contraceptive measures; Serum pregnancy test must be negative within 7 days before the experimental drug for women of childbearing age.

Exclusion Criteria:

-

Participants with mild to moderate liver impairment who meet any of the following criteria will not be eligible for this study:

* Subjects had any of the following conditions: drug-induced liver injury; history of liver transplantation; liver failure, or cirrhosis with grade 3/4 hepatic encephalopathy, esophageal and gastric varices bleeding and other complications considered inappropriate by researchers; severe / advanced peritoneal effusion or pleural effusion requiring puncture drainage and albumin supplement; patients with hepatorenal syndrome; patients with hepatorenal syndrome;
* Biliary cirrhosis, biliary obstruction, cholestatic liver disease and other diseases that affect bile excretion;
* Patients with severe portal hypertension or previous portosystemic shunt, including transjugular intrahepatic portosystemic shunt;
* In addition to primary liver diseases, those who had previously suffered from serious primary diseases of other important organs were not suitable for the trial according to the judgment of the researchers;
* Any of the following conditions occurred within 6 months prior to the study: Myocardial infarction, severe / unstable angina, symptomatic congestive heart failure (NYHA class II-IV), supraventricular or ventricular arrhythmias;
* History of malignant tumor in the past 5 years;
* Patients with severe infection, trauma, gastrointestinal surgery or other major surgical operations within 4 weeks before screening;
* History of drug use, or have a history of drug abuse in the past five years, or have a positive drug screening (except those with drug screening positive due to concomitant drug use);
* HIVAb positive, syphilisAb positive;
* Pregnant or lactating women;
* Strong inducers or inhibitors of CYP3A4, CYP2C9 or CYP2C8 were taken within 14 days before administration of the study drug; used traditional Chinese medicine, dietary supplements and vitamins;
* Subjects with other factors not suitable to participate in this study were considered by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day1~Day9
  Maximum concentration
AUC0-t | Day1~Day9
  Area under the concentration time curve from time zero to time t
AUC0-∞ | Day1~Day9
  Area under the concentration time curve extrapolated to infinity

IPD SHARING:
Plan to Share IPD: No